CLINICAL TRIAL: NCT00003749
Title: A Randomised Trial of Lymphadenectomy and of Adjuvant External Beam Radiotherapy in the Treatment of Endometrial Cancer
Brief Title: Surgery With or Without Lymphadenectomy and Radiation Therapy in Treating Patients With Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066869; MRC-ASTEC; EU-98062
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 1999-04

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; endometrial clear cell carcinoma; endometrial papillary serous carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Chemotherapy, Adjuvant; Brachytherapy; Radiotherapy

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Lymphadenectomy may remove cancer cells that have spread to nearby lymph nodes. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether conventional surgery is more effective with or without lymphadenectomy and/or radiation therapy in treating endometrial cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of conventional surgery with or without lymphadenectomy and/or radiation therapy in treating patients who have endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of conventional surgery alone and conventional surgery plus lymphadenectomy in patients with endometrial cancer preoperatively thought to be confined to the uterine corpus.
* Determine the effect of postoperative adjuvant external beam radiotherapy on quality of life and survival of a subset of these patients at high risk of relapse and with no macroscopic disease after surgery.

OUTLINE: This is a randomized, multicenter study. Patients are randomized in both the surgery and radiotherapy segments of the study.

* Surgery: Patients are randomized to 1 of 2 surgery arms.

  * Arm I: Patients undergo conventional surgery (total abdominal hysterectomy and bilateral salpingo-oophorectomy).
  * Arm II: Patients undergo conventional surgery as in arm I followed by lymphadenectomy with systematic dissection of the iliac and obturator nodes.
* Radiotherapy: Patients at high risk of relapse who have no postoperative macroscopic disease are randomized to 1 of 2 radiotherapy arms. (Patients may enter the radiotherapy randomization after surgery off study.)

  * Arm I: Patients receive in 20-25 fractions of external beam radiotherapy (total dose of 40-46 Gy) over 4-5 weeks.
  * Arm II: Patients receive no external beam radiotherapy. NOTE: Some patients receive vault brachytherapy regardless of radiotherapy randomization.

Quality of life is assessed before therapy and at 2 and 5 years after therapy.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

PROJECTED ACCRUAL: A minimum of 1400 patients will be accrued for the surgical component of this study and at least 900 patients (including additional patients not participating in the surgical component of this study) will be accrued for the radiotherapy component of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Surgical randomization:

* Histologically confirmed endometrial carcinoma
* Disease thought preoperatively to be confined to the uterine corpus

Radiotherapy randomization:

* Must have disease determined postoperatively to be confined to the uterine corpus, irrespective of pelvic node status

  * No cervical stroma invasion (stage IIB)
* Must be macroscopically free of disease (no positive para-aortic nodes)
* Must have high-risk disease defined as one or more of the following:

  * Grade 3 (poorly differentiated)
  * Invasion to the outer half of the myometrium (stage IC)
  * Serous papillary or clear cell type
  * Stage IIA (endocervical glandular involvement)

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior or concurrent malignancy likely to interfere with protocol treatment or comparisons
* Surgical randomization:

  * Must be fit to undergo lymphadenectomy and external beam radiotherapy
* Radiotherapy randomizations:

  * Must be fit to receive external beam radiotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 1998-04; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Amos — Medical Research Council
Locations (3):
- United Kingdom (3):
  - Medical Research Council Clinical Trials Unit, London, England
  - Royal Marsden NHS FoundationTrust - London, London, England
  - St. Mary's Hospital, Manchester, England

REFERENCES:
- [Background] ASTEC/EN.5 Study Group; Blake P, Swart AM, Orton J, Kitchener H, Whelan T, Lukka H, Eisenhauer E, Bacon M, Tu D, Parmar MK, Amos C, Murray C, Qian W. Adjuvant external beam radiotherapy in the treatment of endometrial cancer (MRC ASTEC and NCIC CTG EN.5 randomised trials): pooled trial results, systematic review, and meta-analysis. Lancet. 2009 Jan 10;373(9658):137-46. doi: 10.1016/S0140-6736(08)61767-5. Epub 2008 Dec 16. PMID 19070891
- [Result] Kitchener HC: The effect of incision in the surgical treatment of endometrial cancer and long-term follow-up of a randomized trial of lymphadenectomy: results of the MRC ASTEC trial. [Abstract] J Clin Oncol 29 (Suppl 15): A-e15583, 2011.
- [Result] ASTEC study group; Kitchener H, Swart AM, Qian Q, Amos C, Parmar MK. Efficacy of systematic pelvic lymphadenectomy in endometrial cancer (MRC ASTEC trial): a randomised study. Lancet. 2009 Jan 10;373(9658):125-36. doi: 10.1016/S0140-6736(08)61766-3. Epub 2008 Dec 16. PMID 19070889
- [Result] Barton DP, Naik R, Herod J. Efficacy of systematic pelvic lymphadenectomy in endometrial cancer (MRC ASTEC Trial): a randomized study. Int J Gynecol Cancer. 2009 Nov;19(8):1465. doi: 10.1111/IGC.0b013e3181b89f95. No abstract available. PMID 19893425